CLINICAL TRIAL: NCT05462184
Title: Predictors and Moderators of Effectiveness of Cognitive-Behavioral Therapy and Acceptance and Commitment Therapy in Group Format for Patients With Panic Disorder
Brief Title: Predictors and Moderators of Cognitive-Behavioral Therapy and Acceptance and Commitment Therapy for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Principal Investigator, Leticia León-Quismondo, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAN-MOD
Record Dates: First submitted 2022-06-23; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Panic Disorder; Cognitive-Behavioral Therapy; Acceptance and Commitment Therapy; Predictor
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Active Comparator): CBT followed Craske & Barlow´s (2007) manual, which contains a session-by-session description treatment of panic disorder with CBT. The treatment included the following components: (a) psychoeducation about the nature of anxiety and panic, (b) diaphragmatic breathing training, (c) identification and correction of maladaptive thoughts about anxiety and its consequences, (d) exposure to interoceptive sensations, and (e) exposure to feared situations.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT)
- Acceptance and Commitment Therapy (ACT) (Experimental): ACT was conducted following Eifert & Forsyth´s (2005) manual, which contains a session-by-session description of the application of ACT to anxiety disorders. In the current study, exercises were adapted to the panic disorder treatment. The treatment included the following components: (a) acceptance of internal experiences, (b) cognitive defusion, (c) work with the "self as context", (d) contact with the present moment, (e) work with life values, and values, and (f) commitment to action.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT)
  Arms: Cognitive-Behavioral Therapy (CBT)
Behavioral: Acceptance and Commitment Therapy (ACT)
  Arms: Acceptance and Commitment Therapy (ACT)

SUMMARY:
Objective: Panic disorder is one of the most prevalent anxiety disorders and with the greatest impact on the functionality of patients. Knowing variables that influence the therapies outcome can improve the results of the interventions and reduce the socio-health cost. The current study examined possible predictors and moderators of outcome in cognitive-behavioral therapy (CBT) and acceptance and commitment therapy (ACT). Method: Eighty patients with diagnostic of panic disorder received 12 group sessions of CBT or ACT and were assessed with several measures at baseline, 12 weeks post-treatment and 24 weeks post-treatment.

DETAILED DESCRIPTION:
Panic disorder is characterized by the presence of recurrent and unexpected panic attacks, that is, the person suddenly suffers attacks of intense fear. Panic disorder has a significant prevalence and presents frequent comorbidity with other disorders (anxiety, depression or substance abuse, among others). In addition, its course is usually chronic, leading to a significant functional deterioration for the person, with a deterioration in their quality of life. In addition, it generates high direct and indirect costs (loss of working days, visits to emergency services, medical visits, health expenses, etc.).

The psychological therapy of choice for the treatment of panic disorder is cognitive behavioral therapy (CBT). However, around 25% of patients do not respond successfully to CBT treatment, relapse at the end of therapy or need other additional treatments (Brown & Barlow, 1995; Hofmann et al., 2012). In this context, the study of predictors and moderators of efficacy in psychotherapy is especially relevant, with acceptance and commitment therapy (ACT) being an alternative with growing empirical support. In addition, the group therapy format provides unique qualities and advantages, both at a psychotherapeutic level and in terms of saving resources.

The objective of this study was to analyze the effect of different potentially predictive and moderating variables on the efficacy of cognitive-behavioral therapy and acceptance and commitment therapy in a group format for patients with panic disorder. To this end, a randomized, single-centre, prospective, controlled clinical trial with a 24-week follow-up was carried out.

The sample consisted of 80 patients with panic disorder, randomized into two treatment groups: the experimental group, which received acceptance and commitment therapy, and the active comparator control group, which received cognitive-behavioral therapy. Panic disorder severity was assessed using the Panic Disorder Severity Scale-Self Report (PDSS-SR), fear of physical symptoms using the Body Sensations Questionnaire, BSQ) and the frequency of catastrophic thoughts using the Agoraphobic Cognitions Questionnaire (ACQ). These three measurements were taken before and at the end of treatment, as well as at three months of follow-up.

The potential predictors and moderators analyzed were age, gender, duration of the disorder, motivation to change using the University of Rhode Island Change Assessment Scale (URICA), responsibility through the Five Factor Personality Inventory (Neo Five Factor Inventory, NEO-FFI) and experiential avoidance with the Acceptance and Action Questionnaire-II (AAQ-II).

Participants were randomized to the two treatment groups (CBT or ACT). In both groups, the patients received 12 therapy sessions of 1 hour and 30 minutes duration, with a weekly frequency.

Data analysis was performed using the statistical computing software R version 3.5 and its random forest and Ime4 packages. Statistical analysis was performed by intention to treat (ITT). For the comparison of the sociodemographic and clinical characteristics between the two groups, the Student's t-test was used for the quantitative variables and the Chi-square test for the qualitative variables. To test the hypotheses, a model was designed to perform the analysis of covariance (ANCOVA) type III, which incorporates interactions, considering the time factor of the treatments as a covariate. Post-hoc analyzes were performed with the multcomp package built into the R statistical computing software, which allows performing Tukey-type simultaneous comparison tests for generalized models and generalized mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Panic Disorder diagnostic DSM-5.
* Between 18 and 65 years of age.
* Medication-free or no change in the last month.
* Not undergoing other psychotherapy.

Exclusion Criteria:

* Primary diagnosis of a disorder other than panic disorder.
* Active suicidal ideation.
* Substance abuse or dependence.
* Cognitive impairment, neurological disorders or intellectual disability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline level of Severity of Panic Disorder at 12 weeks and 24 weeks post-treatment. | Baseline, 12 weeks post-treatment and 24 weeks post-treatment.
  It is evaluated through the Panic Disorder Severity Scale-Self Report. It is a self-administered scale whose objective is to determine the level of severity of panic disorder in the last month. It is composed of 7 items, which explore: (1) frequency of panic attacks, (2) distress provoked by panic attacks, (3) anticipatory anxiety, (4) agoraphobic fear and avoidance, (5) fear and/or avoidance of situations, (6) impairment and/or interference in work activity, and (7) impairment and/or interference in social activity. The patient answers using a Likert-type scale from 0 to 4, with 0 being the minimum and 4 the maximum severity of symptoms. It provides a profile of the intensity and presence of symptoms in the last month.
Change from Baseline degree of Fear of Physical Symptoms at 12 weeks and 24 weeks post-treatment. | Baseline, 12 weeks post-treatment and 24 weeks post-treatment.
  It is evaluated through the Body Sensations Questionnaire. It is a self-administered questionnaire composed of 17 items plus 1 final open-ended item. The subject responds to each item according to a 5-point Likert-type scale. This questionnaire evaluates the degree of fear or concern generated by each of the physical symptoms that occur during panic attacks. The final score is obtained by calculating the mean of the 17 items. A high score is indicative of a great fear of the physical symptoms.
Change from Baseline frequency of Agoraphobic Cognitions at 12 weeks and 24 weeks post-treatment. | Baseline, 12 weeks post-treatment and 24 weeks post-treatment.
  It is evaluated through the Agoraphobic Cognitions Questionnaire. It is a self-administered questionnaire composed of 14 items (plus a final open-ended item) on a 5-point Likert-type scale. It evaluates the frequency with which the patient has catastrophic thoughts about the negative consequences of experiencing anxiety when anxious. It is composed of two subscales: catastrophic thoughts about physical consequences of anxiety (heart attack, tumor, etc.) and catastrophic thoughts about social and behavioral consequences (making a fool of oneself, going crazy, etc.). An overall score is obtained by calculating the mean of the total items and the scores on the two subscales: physical level and social-behavioral level.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia León-Quismondo, Principal Investigator — University of Alcala
Locations (1):
- Príncipe de Asturias University Hospital, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice guideline for the treatment of patients with panic disorder. Work Group on Panic Disorder. American Psychiatric Association. Am J Psychiatry. 1998 May;155(5 Suppl):1-34. No abstract available. PMID 9585731
- [Background] Andlin-Sobocki P, Wittchen HU. Cost of anxiety disorders in Europe. Eur J Neurol. 2005 Jun;12 Suppl 1:39-44. doi: 10.1111/j.1468-1331.2005.01196.x. No abstract available. PMID 15877777
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Craske MG, Niles AN, Burklund LJ, Wolitzky-Taylor KB, Vilardaga JC, Arch JJ, Saxbe DE, Lieberman MD. Randomized controlled trial of cognitive behavioral therapy and acceptance and commitment therapy for social phobia: outcomes and moderators. J Consult Clin Psychol. 2014 Dec;82(6):1034-48. doi: 10.1037/a0037212. Epub 2014 Jul 7. PMID 24999670
- [Background] Gloster AT, Sonntag R, Hoyer J, Meyer AH, Heinze S, Strohle A, Eifert G, Wittchen HU. Treating Treatment-Resistant Patients with Panic Disorder and Agoraphobia Using Psychotherapy: A Randomized Controlled Switching Trial. Psychother Psychosom. 2015;84(2):100-109. doi: 10.1159/000370162. Epub 2015 Feb 21. PMID 25722042
- [Background] Niles AN, Wolitzky-Taylor KB, Arch JJ, Craske MG. Applying a novel statistical method to advance the personalized treatment of anxiety disorders: A composite moderator of comparative drop-out from CBT and ACT. Behav Res Ther. 2017 Apr;91:13-23. doi: 10.1016/j.brat.2017.01.001. Epub 2017 Jan 4. PMID 28110111
- [Background] Wolitzky-Taylor KB, Arch JJ, Rosenfield D, Craske MG. Moderators and non-specific predictors of treatment outcome for anxiety disorders: a comparison of cognitive behavioral therapy to acceptance and commitment therapy. J Consult Clin Psychol. 2012 Oct;80(5):786-99. doi: 10.1037/a0029418. Epub 2012 Jul 23. PMID 22823858